CLINICAL TRIAL: NCT01000636
Title: Gene Expression in Renal Transplant Patients With Field Actinic Keratosis Undergoing Metvix® PDT
Brief Title: Gene Expression in Renal Transplant Patients With Field Actinic Keratosis Undergoing Metvix® Photodynamic Therapy (PDT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RD.03.SPR.29061; Eudract # :2008-001603-30
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Actinic Keratosis
Keywords: Renal transplant patients; Actinic Keratoses; Metvix PDT; Field cancerisation; Gene expression
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metvix PDT (Experimental)
  Interventions: Procedure: Metvix PDT

INTERVENTIONS:
Procedure: Metvix PDT — Methyl aminolevulinate cream will be applied for 3 hours on the whole target field.
  The target field will then be exposed to red light using Aktilite 128 lamp.

SUMMARY:
The aim of this study is to determine possible molecular changes on large scale gene expression profiling after treatment with Metvix photodynamic therapy (PDT) of actinic keratoses (AK) and cancerised field in renal transplant recipients.

DETAILED DESCRIPTION:
In this study, the whole target area defined by the investigator will be treated by Metvix PDT: this means that both lesions and sub-clinical lesions will be exposed to Metvix PDT. Biopsies will be performed in both regions: lesional and peri-lesional ones. This will allow us to compare pre and post treatment molecular changes that occurred in these regions and so to evaluate if Metvix PDT acts on the sub-clinical lesions.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant with an history of immunosuppression from 5 to 15 years,
* Presenting at least 4 discrete AK lesions, mild or moderate, either on the face, the scalp, forearms or the chest.

Exclusion Criteria:

* At risk in terms of precautions, warnings, and contra-indication referred in the package insert of Metvix®,
* AK lesions clinically atypical or suspicious for malignancy on the target field,
* Any of the following topical treatments within the specified washout period at Screening:

  * 5-FU, Imiquimod, Diclofenac sodium: 3 months,
  * Cryotherapy: 3 months,
  * PDT: 3 months,
  * Other less common AK treatments: 3 months.
* Systemic retinoids within the last month prior to Screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John T. Lear, MB,Ch.B,M.D, Principal Investigator — Manchester Royal Infirmary
Locations (1):
- Department of Dermatology of Manchester Royal Infirmary, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 subjects have been enrolled in one site at United Kingdom. First subject included on: March 11th 2010; Last subject out: October 7th 2011
Period: Overall Study
Arm/Group | Metvix® Photodynamic Therapy (PDT)
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Only 9 subjects out of 10 planned ones by the protocol have been included
Arm/Group | Metvix PDT
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lesion Count at Week 18
Description: Percent Change in Lesion Counts at Week 18: Week 18 count minus Baseline count divided by Baseline count multiplied by 100.
Time Frame: Baseline and Week 18.
Population: This trial was of exploratory nature, no statistical rationale for sample size exists. Analysis was performed on Intent to treat (ITT) population that consisted of the entire population enrolled and randomized (i.e., assigned a treatment number). Here, "Overall Number of Participants Analyzed" = participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metvix® Photodynamic Therapy (PDT)
Number analyzed (Participants) | 8
percent change | 95.5 (9.1)

2. Secondary Outcome: Global Percent Change From Baseline in AK Lesion Count in the Target Field (Including New and Recurrent Lesions) at Month15
Time Frame: Baseline and Month15
Population: This trial is of exploratory nature, no statistical rationale for sample size exists. This population consists of the entire population enrolled and randomized (i.e., assigned a treatment number).
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Metvix® Photodynamic Therapy (PDT)
Number analyzed (Participants) | 9
Percent change from baseline | 71 (41.4)

ADVERSE EVENTS:
Time Frame: From Screening visit up to Month 15/early termination visit
Description: Questioning of subjects at each follow up visit
Arm/Group | Metvix® Photodynamic Therapy (PDT)
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix® Photodynamic Therapy (PDT) (N=9)
Urinary Track Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix® Photodynamic Therapy (PDT) (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Application site pain (General disorders) | 2 (2)
Influenza Like illiness (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Migraine (Nervous system disorders) | 1 (1)
Erectile dysfuntion (Reproductive system and breast disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 5 (10)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitation or caveat on this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide his draft of such publication to sponsor to review and approve at least 2 months prior to the date of intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.